CLINICAL TRIAL: NCT02479425
Title: Two Pints Versus Three Points Turning in Prevention of Bed Sores in Critically Ill Patients
Brief Title: Two Points Versus Three Points Turning in Prevention of Bed Sores in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Ahmed M El-Mehalawy, Ahmed M El-Mehalawy, MD, lecturer of Critical Care Medicine, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Faculty of Medicine 09052011
Record Dates: First submitted 2015-06-10; First posted 2015-06-24 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Pressure Ulcer
Keywords: pressure ulcer; Positioning
MeSH Terms: conditions — Pressure Ulcer | interventions — Patient Positioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 point turning (Active Comparator): patients nursed by the traditional re-positioning (two hours on back, two hours on right and two hours on left).
  Interventions: Procedure: patient positioning
- 2 points turning (Experimental): patients nursed on the right and left side sonly in 30ْ avoiding the back
  Interventions: Procedure: patient positioning

INTERVENTIONS:
Procedure: patient positioning — positioning patients, every 2 hours, either to standard (right, back, left sides) or only to right and left sides

SUMMARY:
Several studies were searched the preventive measures of bed sores. Although repositioning is the mainstay in most preventive measures, there is no evidence to recommend specific turning regimen.

The aim of this study is to comparative the impact of the two points repositioning in lateral lying position on the right and left versus the traditional three points repositioning on the right, back, and left in the occurrence of bed sores.

This study was conducted on 150 patients admitted to the critical care department of Alexandria Main University Hospital after obtaining an informed consent from their relatives.

The investigators excluded patients who: have active or healed bed sores.

Patients were randomly divided into two groups by allocated randomization:

* Group 1: traditional three points rotation.
* Group 2: two points rotation.

DETAILED DESCRIPTION:
Several studies were searched the preventive measures of bed sores. Although repositioning is the mainstay in most preventive measures, there is no evidence to recommend specific turning regimen.

Aim of the study:

The aim of this study was designed to evaluate the comparative impact of the two points repositioning in lateral lying position on the right and left versus the traditional three points repositioning on the right, back, and left in the occurrence of bed sores.

Patients:

This study was conducted on 150 patients admitted to the critical care department of Alexandria Main University Hospital after obtaining an informed consent from their relatives.

The investigators excluded patients who: have active or healed bed sores.

Patients were randomly divided into two groups by allocated randomization:

* Group 1: traditional three points rotation.
* Group 2: two points rotation.

Methods:

The studied patients were subjected to:

Complete history taking, physical examination, primary ICU diagnosis, routine laboratory investigation and recording Glasgaw coma scale (GCS), use of sedation, vasopressors and mechanical ventilation

Patients in group 1 nursed by traditional protocol [ two hours on the right side in 30 degree lateral position, two hours on the back and two hours on the left side in 30 degree lateral position] Patients in group 2 nursed in lateral position with 30 degree two hours on the right and two hours on the left with elevation of the head of bed by 30 degree in the two groups.

both groups were monitored for bed sores incidence, timing and sites of occurence

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to critical care medicine department and expected to have long stay

Exclusion Criteria:

* active or healed bed sores

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
pressure ulcer occurence | 21 days
  incidence